CLINICAL TRIAL: NCT02152774
Title: A Prospective Study to Assess the Hypotensive Efficacy of Rho-Kinase Inhibitor AR-12286 Ophthalmic Solution 0.5% and 0.7% in Patients With Chronic Angle-closure Glaucoma
Brief Title: A Study to Assess the Effect of Rho-Kinase Inhibitor AR-12286 Ophthalmic Solution 0.5% and 0.7% in Patients With Chronic Angle-closure Glaucoma
Acronym: ROCK - CACG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New York Glaucoma Research Institute (Other)
Responsible Party: Principal Investigator, Jessica Jasien, Co-Investigator, New York Glaucoma Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14.12
Record Dates: First submitted 2014-05-23; First posted 2014-06-02 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Angle-closure Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 0.5% Rho-Kinase Inhibitor (Experimental): AR-12286 is a novel, potent Rho-kinase inhibitor developed by Aerie Pharmaceuticals, Inc., Bridgewater, NJ. It has single-digit nanomolar inhibitory activity against Rho-kinase in enzymatic inhibition assays. Mechanism-of action studies in monkeys demonstrate that AR-12286 lowers IOP primarily by increasing aqueous humor outflow through the trabecular meshwork Rho-kinase AR-12286 is well tolerated and produces clinically and statistically significant ocular hypotensive efficacy in patients with ocular hypertension and glaucoma. It is well tolerated by most patients and the only side effect was ocular hyperemia in a minority of subjects. It is currently in phase II testing.
  Interventions: Drug: Rho-Kinase Inhibitor
- 0.7% Rho-Kinase Inhibitor (Experimental): AR-12286 is a novel, potent Rho-kinase inhibitor developed by Aerie Pharmaceuticals, Inc., Bridgewater, NJ. It has single-digit nanomolar inhibitory activity against Rho-kinase in enzymatic inhibition assays. Mechanism-of action studies in monkeys demonstrate that AR-12286 lowers IOP primarily by increasing aqueous humor outflow through the trabecular meshwork Rho-kinase AR-12286 is well tolerated and produces clinically and statistically significant ocular hypotensive efficacy in patients with ocular hypertension and glaucoma. It is well tolerated by most patients and the only side effect was ocular hyperemia in a minority of subjects. It is currently in phase II testing.
  Interventions: Drug: Rho-Kinase Inhibitor

INTERVENTIONS:
Drug: Rho-Kinase Inhibitor

SUMMARY:
To evaluate the ocular hypotensive efficacy of Rho kinase Inhibitor (AR-12286 0.5% and 0.7%) ophthalmic solutions in patients diagnosed with chronic angle-closure glaucoma treated for 6 months.

Secondary Outcome

Secondary objectives are:

1. To evaluate the early effect of Rho kinase Inhibitor (AR-12286) in reducing intraocular pressure (IOP).
2. To evaluate the long term effect of the drug on IOP.
3. To determine if AR-12286 can be used as directed therapy for CACG, reducing or eliminating the structural blockage of the trabecular meshwork that leads to development of elevated IOP.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 50 and 85 years old; of either sex.
2. Patients with CACG with ≥180⁰ PAS
3. IOP ≥22 mmHg prior to initiation of treatment in one or both eyes with two measurements taken two hours apart
4. No previous intraocular surgery except clear cornea phacoemulsification.
5. Corrected visual acuity in both eyes ≥20/50 in the eligible eye
6. Not more than 6 diopters spherical equivalent on the study eye
7. Not more than 3 diopters cylinder equivalent on the study eye
8. Have given written informed consent, prior to any investigational procedures.
9. Ability to attend for the 6-month duration of the study

Exclusion Criteria:

1. Open angle glaucoma
2. Closed angle glaucoma with <180⁰ PAS
3. Intraocular pressure >35 mmHg
4. Severe glaucomatous damage
5. Known hypersensitivity to any component of the formulation (benzalkonium chloride, etc.), or to topical anesthetics.
6. Previous intraocular surgery except clear cornea phacoemulsification.
7. Clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study.
8. Ocular medication of any kind within 30 days of base-line visit, with the exception of ocular hypotensive medications and/or drops for treatment of dry eye syndrome (which may be used throughout the study).
9. Any abnormality preventing reliable applanation tonometry of either eye.
10. Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, endocrine or cardiovascular disorders) which might interfere with the study.
11. Changes of systemic medication that could have a substantial effect on IOP anticipated during the study.
12. Participation in any investigational study within the past 30 days.
13. Inability to perform reliable VF testing.
14. Unwilling to sign the consent form approved by the Institutional Review Board (IRB) of the New York Eye and Ear Infirmary.
15. Self-reported poor compliance to treatment.
16. Reluctance to return for scheduled follow-up visits.
17. Patients not able to understand the nature of the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Long Lasting effect of study drug to reduce IOP | 6 Months
  To evaluate the ocular hypotensive efficacy of Rho kinase Inhibitor (AR-12286 0.5% and 0.7%) ophthalmic solutions in patients diagnosed with CACG treated for 6 months.

SECONDARY OUTCOMES:
Secondary Outcome | 6 Months
  To determine if AR-12286 can be used as directed therapy for CACG, reducing or eliminating the structural blockage of the trabecular meshwork that leads to development of elevated IOP.

CONTACTS AND LOCATIONS:
Locations (1):
- Glaucoma Associates of New York, New York, New York, United States